CLINICAL TRIAL: NCT03378635
Title: A Phase 3, Randomized, Double-blind, Parallel Trial to Confirm the Clinical Efficacy and Safety of Dasiglucagon in Rescue Treatment of Hypoglycemia in Subjects With Type 1 Diabetes Mellitus Compared to Placebo and With Reference to GlucaGen
Brief Title: A Trial to Confirm the Efficacy and Safety of Dasiglucagon in the Treatment of Hypoglycemia in Type 1 Diabetes Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-16137
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
Keywords: Dasiglucagon; Glucagon analog
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1 | interventions — dasiglucagon; Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dasiglucagon (Experimental): Single fixed dose (s.c.injection) of dasiglucagon
  Interventions: Drug: Dasiglucagon
- Placebo (Placebo Comparator): Single fixed dose (s.c.injection) of placebo
  Interventions: Drug: Placebo
- GlucaGen® (Active Comparator): Single fixed dose (s.c.injection) of GlucaGen®
  Interventions: Drug: GlucaGen

INTERVENTIONS:
Drug: Dasiglucagon — Glucagon analog
  Other Names: ZP4207
  Arms: Dasiglucagon
Drug: GlucaGen — Native glucagon
  Other Names: GlucaGen HypoKit
  Arms: GlucaGen®
Drug: Placebo — Placebo for dasiglucagon
  Other Names: Placebo for dasiglucagon
  Arms: Placebo

SUMMARY:
The objective of the trial is to demonstrate superiority of dasiglucagon compared to placebo following a single subcutaneous dose administered to subjects with type 1 diabetes mellitus (T1DM) with insulin-induced hypoglycemia. Additionally to compare the glycemic response observed after administration dasiglucagon with that of GlucaGen®.

DETAILED DESCRIPTION:
This was a global, multicenter, randomized, parallel, and double-blind clinical trial confirming the efficacy and safety of dasiglucagon for insulin-induced hypoglycemia in patients with T1DM. The patients were randomized 2:1:1 to receive a single subcutaneous 0.6 mg dose of dasiglucagon, placebo, or a 1 mg dose of GlucaGen and followed for at least 28 days after receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects with type 1 diabetes mellitus (T1DM) for at least 1 year, diagnostic criteria as defined by the American Diabetes Association
* Treated with insulin for T1DM for at least 1 year and with stable insulin treatment (defined as no more than a 10-unit daily variation in total daily insulin dose) 30 days prior to screening
* Hemoglobin A1c <10%

Exclusion Criteria:

* Previously treated with dasiglucagon (previously referred to as ZP4207)
* Known or suspected allergy to trial product(s) or related products
* Females who are pregnant according to a positive pregnancy test, are actively attempting to get pregnant, or are lactating.
* History of hypoglycemic events associated with seizures in the last year prior to screening
* History of severe hypoglycemia in the last month prior to screening
* Active malignancy within the last 5 years
* Current bleeding disorder, including anti-coagulant treatment
* Known presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma (i.e. insulin secreting pancreas tumor)
* Use of a daily systemic beta-blocker drug, indomethacin, warfarin or anticholinergic drugs in the previous 28 days before Day 1 of this trial
* Clinically significant abnormal ECG at screening as judged by the investigator
* Donation of blood or plasma in the past month, or in excess of 500 mL within 12 weeks prior to screening
* Surgery or trauma with significant blood loss within the last 2 months prior to screening
* A positive result in the alcohol and/or urine drug screen at the screening visit. Significant history of alcoholism or drug abuse as judged by the investigator or consuming more than 24 g alcohol per day for men, or more than 12 g alcohol per day for women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Sylvest, MSc Pharm, Study Director — Zealand Pharma
Locations (5):
- ProSciento, Chula Vista, California, United States
- Clinical Research Center, Medizinische Universität Graz, Graz, Austria
- LMC Diabetes & Manna Research, Toronto, Canada
- Germany (2):
  - Profil, Mainz
  - Profil, Neuss

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pieber TR, Aronson R, Hovelmann U, Willard J, Plum-Morschel L, Knudsen KM, Bandak B, Tehranchi R. Dasiglucagon-A Next-Generation Glucagon Analog for Rapid and Effective Treatment of Severe Hypoglycemia: Results of Phase 3 Randomized Double-Blind Clinical Trial. Diabetes Care. 2021 Jun 1;44(6):1361-1367. doi: 10.2337/dc20-2995. PMID 35239971

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasiglucagon 0.6 mg: Single fixed dose (s.c.injection) of dasiglucagon
  Dasiglucagon: Glucagon analog
- GlucaGen® 1.0 mg: Single fixed dose (s.c.injection) of GlucaGen®
  GlucaGen: Native glucagon
Period: Overall Study
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Started (Started is defined as randomized) | 84 | 43 | 43
Randomized and Exposed to Treatment | 82 | 43 | 43
Completed | 82 | 43 | 43
Not Completed | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg | Total
Number analyzed (Participants) | 82 | 43 | 43 | 168
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.1) | 38.0 (13.1) | 40.2 (11.5) | 39.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 16 | 15 | 63
  Male | 50 | 27 | 28 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 80 | 41 | 40 | 161
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 1 | 2 | 4
  White | 76 | 39 | 39 | 154
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 10 | 10 | 38
  Austria | 33 | 0 | 0 | 33
  United States | 12 | 6 | 6 | 24
  Germany | 19 | 27 | 27 | 73

OUTCOME MEASURES:

1. Primary Outcome: Time to Plasma Glucose Recovery
Description: Plasma glucose recovery is defined as first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline without administration of rescue intravenous glucose. The outcome measure used a Kaplan-Meier estimate with 95% confidence interval. Treatment groups without censoring utilized a distribution free method to compute the confidence interval for median time.
Time Frame: 0-45 minutes after dosing
Population: Full analysis set of all randomized patients who received at least one dose of trial product
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
minutes | 10 [10 to 10] | 40 [30 to 40] | 12 [10 to 12]
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The treatment group difference between dasiglucagon and placebo was evaluated inferentially using a pairwise two-sided log rank test. Kaplan-Meier estimate with 95% CI, p-value based on treatment group difference between dasiglucagon and placebo using a two-sided log-rank test stratified by injection site. Treatment groups without censoring utilized a distribution free method to compute the confidence interval for median time; Test type: Superiority; p < 0.001, Log Rank

2. Secondary Outcome: Plasma Glucose Recovery
Description: Plasma glucose recovery within 30 minutes, within 20 minutes, within 15 minutes, and within 10 minutes after study drug injection without administration of rescue IV glucose. Plasma glucose recovery was defined as the first increase in plasma glucose of ≥20 mg/dL (1.1 mmol/L) from baseline without administration of rescue intravenous glucose.
Time Frame: 0-30 minutes after dosing: assessed at 10, 15, 20 and 30 minutes after study drug injection
Population: Full analysis set of all randomized patients who received at least one dose of trial product
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
Participants
  Glucose recovery at 30 minutes | 82 | 20 | 43
  Glucose recovery at 20 minutes | 81 | 6 | 42
  Glucose recovery at 15 minutes | 81 | 1 | 41
  Glucose recovery at 10 minutes | 53 | 0 | 21
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Pairwise test of independent binomial proportions with Fisher's Exact test comparing dasiglucagon versus placebo. Testing followed an a priori defined hierarchical inferential test order, proceeding until the first failure to reject the null hypothesis comparing dasiglucagon versus placebo; Test type: Superiority; p < 0.001, Fisher Exact — p-value was <0.001 at all time points (10, 15, 20 and 30 minutes)

3. Secondary Outcome: Plasma Glucose Changes From Baseline
Description: Plasma glucose changes from baseline at 30 minutes, 20 minutes, 15 minutes and 10 minutes after study drug injection without administration of rescue intravenous glucose
Time Frame: 0-30 minutes after dosing: assessed at 10, 15, 20 and 30 minutes after study drug injection
Population: Full analysis set of all randomized patients who received at least one dose of trial product
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
mg/dL
  At 30 minutes | 90.9 (18.2) | 19.1 (13.0) | 88.5 (19.2)
  At 20 minutes | 59.7 (15.0) | 8.7 (10.8) | 58.4 (15.6)
  At 15 minutes | 43.5 (12.51) | 6.65 (6.82) | 44.1 (14.0)
  At 10 minutes | 23.9 (9.84) | -0.14 (5.65) | 22.0 (10.0)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; Plasma glucose (PG) change from baseline at rescue was carried forward in patients who required rescue intravenous (IV) glucose before reaching PG recovery. Change from baseline was analyzed using an ANCOVA, with treatment group as fixed effect and baseline PG as covariate. Group difference was evaluated inferentially following an a priori defined hierarchical test order, proceeding until the first failure to reject the null hypothesis; Test type: Superiority; p < 0.001, ANCOVA — The p-value was <0.001 at all time points (10, 15, 20 and 30 minutes)

4. Secondary Outcome: Time to Target
Description: Time to first plasma glucose concentration ≥70 mg/dL (3.9 mmol/L) without administration of rescue intravenous glucose. The outcome measure used a Kaplan-Meier estimate with 95% confidence interval. Treatment groups without censoring utilized a distribution free method to compute the confidence interval for median time.
Time Frame: 0-45 minutes after dosing
Population: Full analysis set of all randomized patients who received at least one dose of trial product
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
minutes | 8 [8 to 8] | 25 [20 to 30] | 8 [8 to 10]
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The treatment group difference between dasiglucagon and placebo was evaluated using a Kaplan-Meier estimate with 95% confidence interval, p-value based on a pairwise two-sided log-rank test versus placebo; Test type: Superiority; p < 0.001, Log Rank

5. Secondary Outcome: Pharmacodynamics - Area Under the Effect Curve
Description: Plasma glucose response as area under the effect curve (AUE) above baseline from time zero to 30 minutes. Samples were collected pre-dose, and at 4, 6, 8, 10, 12, 15, 17, 20, 25 and 30 minutes after dosing.
Time Frame: 0-30 minutes after dosing
Population: Full analysis set of all randomized patients who received at least one dose of trial product
Measure: Mean (Standard Deviation); unit: mg*h/dL
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
mg*h/dL | 21.0 (5.26) | 3.57 (2.86) | 20.4 (5.49)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs Placebo; The log-transformed AUC endpoint was analyzed using an analysis of covariance model with treatment as fixed effect and baseline plasma glucose modeled as a covariate. The least squares means treatment group differences were back-transformed (anti-logged) for presentation as a ratio of the treatment group geometric means, with their corresponding 95% confidence interval; Test type: Superiority; p < 0.001, ANCOVA; Mean Difference (Net) = 0.131, 95% CI 2-sided [0.1 to 0.171]

6. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the drug concentration curve from time zero to 90 minutes, AUC0-90min. To calculate the AUC the standard trapezoidal method was used, based on actual rather than nominal time points. Samples were collected pre-dose, and at 15, 30, 35, 40, 50, 60, 90 and 120 minutes after dosing.
Time Frame: 0-90 minutes after dosing
Population: Full analysis set of all randomized patients who received at least one dose of trial product. No results are presented for the placebo group, as no active drug was given in this group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43
pmol*h/L | 1430 (34.2) | 1300 (27.5)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs GlucaGen® 1.0 mg; Least square mean ratio for GlucaGen: dasiglucagon; Test type: Superiority; p = 0.144, ANCOVA; Mean Difference (Net) = 0.91, 95% CI 2-sided [0.801 to 1.033]

7. Secondary Outcome: Pharmacokinetics - Area Under the Plasma Concentration Curve
Description: Area under the drug concentration curve from time zero to 120 minutes, AUC0-120min. To calculate the AUC the standard trapezoidal method was used, based on actual rather than nominal time points. Samples were collected pre-dose, and at 15, 30, 35, 40, 50, 60, 90 and 120 minutes after dosing.
Time Frame: 0-120 minutes after dosing
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol*h/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43
pmol*h/L | 1770 (31.2) | 1490 (27.2)
Statistical Analysis 1: Comparison: Dasiglucagon 0.6 mg vs GlucaGen® 1.0 mg; Least square mean ratio for GlucaGen: dasiglucagon; Test type: Superiority; p = 0.006, ANCOVA; Mean Difference (Net) = 0.844, 95% CI 2-sided [0.749 to 0.951]

8. Secondary Outcome: Pharmacokinetics - Maximum Plasma Concentration
Description: Maximum plasma drug concentration (Cmax). Maximum plasma drug concentration was determined as the maximum of all valid plasma dasiglucagon/glucagon concentrations. Samples were collected pre-dose, and at 15, 30, 35, 40, 50, 60, 90 and 120 minutes after dosing.
Time Frame: 0-120 minutes after dosing
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43
pmol/L | 1280 (37.7) | 1490 (34.5)

9. Secondary Outcome: Pharmacokinetics - Time to Maximum Plasma Concentration
Description: Time to maximum plasma drug concentration (tmax). Median Tmax was determined as the time point where the maximum of all valid plasma dasiglucagon/glucagon concentration measurements for each measurement series was observed. Samples were collected pre-dose, and at 15, 30, 35, 40, 50, 60, 90 and 120 minutes after dosing.
Time Frame: 0-120 minutes after dosing
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43
hours | 0.670 [0.250 to 1.00] | 0.250 [0.230 to 0.670]

10. Secondary Outcome: Immunogenicity - Occurence of Anti-drug Antibodies
Description: Occurence of antibodies against dasiglucagon/GlucaGen
Time Frame: 28 days
Population: The safety analysis set of all randomized patients who received trial medication (which was the same as the full analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43
Participants
  Anti-drug antibodies at follow-up day 28 | 1 | 0
  Anti-drug antibodies at second follow up | 0 | 0

11. Secondary Outcome: Rescue Infusion of IV Glucose During the Hypoglycemic Clamp Procedure
Description: Number of patients receiving administration of rescue infusion of IV glucose during the hypoglycemic clamp procedure. IV = intravenous
Time Frame: 0-45 minutes after dosing
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 82 | 43 | 43
Participants | 0 | 0 | 0

12. Secondary Outcome: Time to First Rescue Infusion of IV Glucose
Description: Time to first rescue administration of rescue infusion of IV glucose. IV = intravenous
Time Frame: 0-45 minutes after dosing
Population: No patients received IV glucose infusions therefore there are no data available for this outcome measure
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the first trial-related activity after the patient had signed the informed consent to the end of the follow-up period, i.e. over 28 days
Description: All AEs, either observed by the investigator or reported by the patient, were recorded by the investigator and evaluated, including diagnosis, if possible. If no diagnosis was made, the investigator was to record each sign and symptom as individual AEs. Information included date and time of onset and resolution, date and time of investigator's first information on the AE, seriousness, severity, casual relationship with investigational product, interruption/withdrawal of treatment and outcome.
Arm/Group | Dasiglucagon 0.6 mg | Placebo | GlucaGen® 1.0 mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 66/82 | 14/43 | 32/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasiglucagon 0.6 mg (N=82) | Placebo (N=43) | GlucaGen® 1.0 mg (N=43)
Headache (Nervous system disorders) | 10 (10) | 2 (2) | 5 (5)
Nausea (Gastrointestinal disorders) | 45 (46) | 1 (1) | 23 (24)
Vomiting (Gastrointestinal disorders) | 19 (25) | 1 (1) | 9 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 23 (39) | 5 (6) | 9 (10)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 2 (2) | 2 (2)
Injection site edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03378635/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT03378635/SAP_001.pdf